CLINICAL TRIAL: NCT05925725
Title: Clinical Efficacy and Safety of Loxacon Dietary Supplement Capsules at the Treatment of Patients With Knee Arthrosis. A Multicenter Randomized, Double-blind, Follow-up Clinical Trial
Brief Title: Clinical Efficacy and Safety of Loxacon Dietary Supplement Capsules at Patients With Knee Arthrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Polyclinic of the Hospitaller Brothers of St. John of God, Budapest (Other)
Responsible Party: Principal Investigator, Tamas Bender, professor of Medicine, Polyclinic of the Hospitaller Brothers of St. John of God, Budapest
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: PolyclinicHBSJG physiothetrapy
Record Dates: First submitted 2023-04-07; First posted 2023-06-29 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Osteo Arthritis Knee
Keywords: Boswellia serrata,; Harpagophytum procumbens,; knee OA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Loxacon and Physical Therapy (Active Comparator): physical therapy(exercise) + caps Loxacon
  Interventions: Drug: • harpagozid • boswellin = LOXACON
- Physical therapy and Placebo Loxacon caps (Placebo Comparator): Physical therapy + Placebo caps Loxacon
  Interventions: Drug: • harpagozid • boswellin = LOXACON
- Pphysical therapy(alone) (Active Comparator): Physical therapy
  Interventions: Drug: • harpagozid • boswellin = LOXACON

INTERVENTIONS:
Drug: • harpagozid • boswellin = LOXACON — Exercise therapy
  Other Names: Physiotherapy(exercise)

SUMMARY:
The study will be a multicenter, randomized, double-blind, follow-up clinical trial.

Neither the examining doctor nor the patient knows which capsule they will receive. Just the test unlock the codes after completion. T

DETAILED DESCRIPTION:
The study will be a multicenter, randomized, double-blind, follow-up clinical trial.

Neither the examining doctor nor the patient knows which capsule they will receive. Just the test unlock the codes after completion. The randomization was performed externally, not included in the study performed by a person. Number of patients: a total of 105 patients / 25-25 per clinic (with 8 patients each in three treatment groups) Three treatment groups

* 35 people physical therapy + Loxacon
* 35 main physical therapy + Placebo
* 35 people only for physical therapy Physiotherapy(exercise) takes place according to a uniform protocol. Physiotherapy 2x30 minutes per week for 5 weeks (10 times in total). The course of the investigation

  1. st visit: selection, filling in questionnaires
  2. nd visit: after the 10th exercise session, while taking Loxacon/placebo, filling in questionnaires
  3. rd visit: Uniformly after another 2 months of taking Loxacon, in all three groups, completing questionnaires After the first 5 weeks, all three branches will receive enough Loxacon capsules for 2 months! The parameters to be tested

     * WOMAC test
     * VAS
     * EQ-5D-5L quality of life test
     * Goniometer angle measurement The test is completed by patients who participated in more than 70% of the treatment! Monitoring of side effects It is the duty of the doctor of the given center - who reports to the investigator.

ELIGIBILITY:
Inclusion Criteria Must be able to swallow tablets

* According to the ACR (American College of Rheumatology) knee arthrosis criteria, knee arthrosis supported by an imaging procedure (comparative knee X-ray). Both in the case of knee involvement, the more complaining knee will be examined! 2. A patient reporting knee pain characteristic of knee arthrosis for at least 3 months, where the VAS value 40-70 mm. 3. With a diagnosis of mild and moderate knee arthrosis. 4. Male or female patients between the ages of 40 and 80. 5. With a BodyMassIndex between 25-35.

Exclusion Criteria:EXCLUSION CRITERIA

* Intra-articular corticosteroid within 3 months before starting treatment injection.
* Intra-articular hyaluronic acid treatment within 6 months or such treatment during the examination treatment.
* Physiotherapy treatment received within 3 months prior to the start of the treatment.
* NSAID changed within 3 months prior to treatment or during treatment, or chondroprotective treatment.
* In inflammatory rheumatological diseases (RA, SPA, APs, crystal arthropathies, etc.) suffering patient.
* Knee surgery within 6 months prior to the examination.
* Presence of a metal implant in the knee joint.
* Patients who had a knee joint injury within 6 months prior to the examination.
* Patients with a palpable fluid collection in the knee or Baker's cyst.
* Uncooperative patients, patients with inadequate mental or psychological status.

Clinical diagnosis of Alzheimer's Disease

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | one year
  The test questions are scored on a scale of 0-4, whichcorrespondto: None (0), Mild (1)
  , Moderate (2), Severe (3), and Extreme (4).
Visual analog The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be') | "through study completion, an average of 1 year".
  pain measurement The higher score the worser
GONIOMETER | "through study completion, an average of 1 year".
  Range of motion(0-140)Goniometry is the art and science of measuring the joint ranges in each plane of the joint.The hihger the movements's degree the better the result of exercise
Knee Injury and Osteoarthritis Outcome Score (KOOS) | "through study completion, an average of 1 year".
  The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, otherSymptoms, Function in dailyliving (ADL), Function in Sport and Recreation (Sport/Rec), and knee-relatedQuality of Life (QOL)KOOS consists of 5 subscales; long-term patient-relevant outcomes following knee injury

SECONDARY OUTCOMES:
Euroquol Group index EQ-5D-he EQ-5D | "through study completion, an average of 1 year".
  is a commonly used general questionnaire belonging to the first group. When filling it out, respondents in 5 dimensions: mobility, self-sufficiency, usual activities, pain/discomfort, anxiety/depression; They can choose from 3 levels (1: least, 3: most).

CONTACTS AND LOCATIONS:
Overall Officials: Zoltán Dégi, M.D, Study Director — Goodwill Pharma; Zoltán Dégi, Study Chair — Goodwill Pharma; Tamas Bender, Principal Investigator — Polyclinic of the Hospitaller Brothers of St. John of God, Budapest
Locations (1):
- Lakitelek foundation, Lakitelek, Hungary

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT05925725/Prot_000.pdf